CLINICAL TRIAL: NCT01388803
Title: Right Side Bronchial Blocker in Video-assisted Thoracoscopic Surgery
Brief Title: The Depth of Right Bronchial Blocker Placement in Taiwanese in Video-assisted Thoracoscopic Surgery(VATS)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ya-Jung Cheng, Department of Anesthesiology, National Taiwan University Hospital
Other Study IDs: 201012143RC
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Lung Tumor; Pneumothorax
Keywords: bronchial blocker; VATS
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective study to demonstrate the optimal depth of right side bronchial blocker for complete right lung separation. Data were collected from all patients who completed right side VATS with right side BB from Jan 2010 through Nov 2010.

DETAILED DESCRIPTION:
After general anesthesia, an 8.0 mm internal-diameter single-lumen endotracheal tube was inserted orally. An independent Coopdech bronchial blocker, which has a formed-curvature near the catheter tip, was directly inserted through the single-lumen endotracheal tube into right main bronchus. Chest inspection, auscultation, fiberoptic bronchoscopy confirmation, if necessary, by visualizing the blocker cuff located at right main bronchus just below the carina was performed firstly. After placing patients in left decubitus position, the position of BB was reconfirmed by auscultation firstly; then complete collapse of the right upper lobe was adjust, if necessary and reconfirmed on the video of thoracoscopy by both surgeon and anesthesiologists. The depth of BB and the need of fiberoptic bronchoscope were recorded. All the patients were extubated in operation room after completion of operation with optimal analgesia. Data collected included; age, sex, body height and weight and the depth of right-sided BB from incisor was then recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving right side VATS( video-assisted thoracoscopic surgery) with right side bronchial blocker

Exclusion Criteria:

* Patients receiving thoracic surgery with double lumen tubes

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving right side VATS( video-assisted thoracoscopic surgery) with right side bronchial blocker
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ya-jung cheng, PhD, Study Director — deaprtment of anesthesiology, national taiwan university hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan